CLINICAL TRIAL: NCT02213692
Title: Comparative Study on Liver Resection Between Harmonic Scalpel Versus Crush-clamping Method: A Prospective Randomized Study
Brief Title: Comparative Study on Liver Resection Between Harmonic Scalpel Versus Crush-clamping Method
Status: Terminated | Type: Observational
Sponsor: Hui-Chuan Sun (Other)
Responsible Party: Sponsor-Investigator, Hui-Chuan Sun, Professor, Fudan University
Organization: Fudan University (Other)
Other Study IDs: D2014-051
Record Dates: First submitted 2014-05-30; First posted 2014-08-11 (Estimated); Last update posted 2016-02-04 (Estimated); Status verified 2016-02

CONDITIONS: Hepatic Neoplasms
Keywords: Liver Resection; Harmonic Scalpel; Crush-clamping; A Prospective Randomized Study
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Crush-clamping Method (group A): Liver parenchymal is crushed by surgeon's fingers or basic surgical clamps to isolate small vessels and biliary radicals, and then divided by suture ligation, electrocautery, or vascular clips.
- Harmonic Scalpel Method (group B): Liver parenchymal transection is transected by harmonic scalpel, and small vessels and biliary radicals (<3mm) is also divided by harmonic scalpel. Vessels and biliary radicals (≥ 3mm) were divided by suture ligation, electrocautery, or vascular clips.

SUMMARY:
Blood loss during liver resection significantly associates with short term operative outcome. The median blood loss during partial liver resection is 700-1200ml in high-volume centers. Conventional method (crush-clamp) has been a standard technique for liver transection. Technique advances related to liver transection have contributed to reduction in blood loss. Several studies have showed that Harmonic Scalpel in liver resection is safe and easy to use. A nonrandomized study showed use of the Harmonic Scalpel was associated with decreased operative time, blood loss and transfusion requirement, and an increased incidence of postoperative bile leakage. However, no randomized study has compared the difference between liver resection using traditional technology and harmonic Scalpel. The objective of this prospective randomized study is to compare the safety and efficacy of liver resection using the harmonic scalpel device with the "crush-clamp" technique in respect to blood loss, liver transection time, hepatic hilum clamping time, hospital stay and postoperative complications.

DETAILED DESCRIPTION:
Blood loss during liver resection significantly associates with short term operative outcome. The median blood loss during partial liver resection is 700-1200ml in high-volume centers. Conventional method (crush-clamp) has been a standard technique for liver transection. Technique advances related to liver transection have contributed to reduction in blood loss. Several studies have showed that Harmonic Scalpel in liver resection is safe and easy to use. A nonrandomized study showed use of the Harmonic Scalpel was associated with decreased operative time, blood loss and transfusion requirement, and an increased incidence of postoperative bile leakage. However, no randomized study has compared the difference between liver resection using traditional technology and harmonic Scalpel. The objective of this prospective randomized study is to compare the safety and efficacy of liver resection using the harmonic scalpel device with the "crush-clamp" technique in respect to blood loss, liver transection time, hepatic hilum clamping time, hospital stay and postoperative complications. All patients submitted to liver resection are randomized into two groups: those submitted to liver resection with the use of "crush-clamp" technique. (group Α) and those with the use of the Harmonic Scalpel device (group Β).

Crush-clamping Method (group A) :Patients submitted to liver resection with the use of "crush-clamping" technique.

Device: Liver parenchymal is crushed by surgeon's fingers or basic surgical clamps to isolate small vessels and biliary radicals, and then divided by suture ligation, electrocautery, or vascular clips.

Harmonic Scalpel (group B) :Patients submitted to liver resection with the use of the Harmonic Scalpel device.Device: liver parenchymal transection is transected by harmonic scalpel, and small vessels and biliary radicals (<3mm) is also divided by harmonic scalpel. Vessels and biliary radicals (≥ 3mm) were divided by suture ligation, electrocautery, or vascular clips.

Primary Outcome Measures:

Blood loss during operation [an expected average of 3 hours] operation][Designated as safety issue: Yes] Postoperative complications including bile leakage, bleeding, morbidity, injured Liver function [Time Frame: participants will be followed for the duration of hospital stay, an expected average of 8 days] [Designated as safety issue: Yes]

Secondary Outcome Measures:

Transection time from Mark of the cutting edge to finish disposed of the cutting edge [Designated as safety issue: No] Hepatic hilar clamping time (Pringle's method) [the duration of clamping of hepatic hilar] [Designated as safety issue: No] Hospital stay [participants will be followed for the duration of hospital stay, an expected average of 8 days] [Designated as safety issue: No] Enrollment: 128 Study Start Date: June 2014 Study Completion Date: May 2015 Primary Completion Date: May 2015 (Final data collection date for primary outcome measure)

Eligibility:

Genders Eligible for Study: Both Accepts Healthy Volunteers: No

Criteria:

Inclusion Criteria:

1. Age ≥18y, and ≤80y;
2. No history of liver resection and radiotherapy
3. Liver function: Child A with a normal prothrombin time (<13 seconds) and international normalized ratio (INR )(<1.15);
4. Extent of resection ≥2 segment or diameter of tumor (single nodule) ≥ 8cm or cumulative diameter of tumor (multiple nodule) ≥ 8cm; Eligible patients will be stratified by resection in left lobe or right lobe.
5. No tumor thrombosis in main trunk or right and left branch of portal vein or major hepatic vein.

Exclusion Criteria:

1. Recurrent liver tumor; or simultaneous resection of other organs except gallbladder
2. Prothrombin time > 13seconds;
3. Blood platelets count (BPC) < 60*109
4. Moderate and severe of esophageal varices detected by CT or MRI
5. Diameter of portal vein > 14mm (color ultrasound)

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18y, and ≤80y;
2. No history of liver resection and radiotherapy
3. Liver function: Child A with a normal prothrombin time (<13 seconds) and INR (1.15);
4. Extent of resection ≥2 segment or diameter of tumor (single nodule) ≥ 8cm or cumulative diameter of tumor (multiple nodule) ≥ 8cm; Eligible patients will be stratified by resection in left lobe or right lobe.
5. No tumor thrombosis in main trunk or right and left branch of portal vein or major hepatic vein.

Exclusion Criteria:

1. Recurrent liver tumor; or simultaneous resection of other organs except gallbladder
2. Prothrombin time > 13S;
3. Blood platelets count (BPC) < 60x109
4. Moderate and severe of esophageal varices detected by CT or MRI
5. Diameter of portal vein > 14mm (color ultrasound)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Genders Eligible for Study: Both Accepts Healthy Volunteers: No
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2014-05; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Blood loss | intraoperatively operation（an average of 3 hours)
  Amount of blood loss will be assayed during operation.

SECONDARY OUTCOMES:
Transection time | from Mark of the cutting edge to finish disposed of the cutting edge (an average of 1 hour)
  Liver transection time from Mark of the cutting edge to finish disposed of the cutting edge will be recorded.
Hepatic hilar clamping time | duration of clamping of hepatic hilar (an average of 30 minutes)
  Hepatic hilar clamping time (Pringle's method) will be recorded.
Hospital stay | dates from admission to discharge (an average of 8 days)
  Time of hospital stay will be recorded.
Postoperative complications | within 7 days after operation
  Postoperative complications including bile leakage, bleeding, morbidity, injured Liver function will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Hui Chuan Sun, Professor, Study Chair — Fudan University; Jia Fan, Professor, Principal Investigator — Fudan University; Jian Zhou, Professor, Principal Investigator — Fudan University; Shuang Jian Qiu, Professor, Principal Investigator — Fudan University; Guo Ming Shi, Asso. Prof., Principal Investigator — Fudan University; Qing Hai Ye, Professor, Principal Investigator — Fudan University; Lu Wang, Professor, Principal Investigator — Fudan University; Xiao Wu Huang, Professor, Principal Investigator — Fudan University; Ning Ren, Professor, Principal Investigator — Fudan University; Jing Xian Yu, Nurse, Principal Investigator — Fudan University; Yang Xu, Asso. Prof., Principal Investigator — Fudan University; Ying Hong Shi, Asso. Prof., Principal Investigator — Fudan University; Xiao Ying Wang, Asso. Prof, Principal Investigator — Fudan University; Jian Sun, Asso. Prof., Principal Investigator — Fudan University; Zheng Wang, Asso. Prof., Principal Investigator — Fudan University; Yong Sheng Xiao, Asso. Prof., Principal Investigator — Fudan University; Pei Chen, Asso. Prof., Principal Investigator — Fudan University; Cheng Huang, Asso. Prof., Principal Investigator — Fudan University; Ying Hao Shen, Asso. Prof., Principal Investigator — Fudan University
Locations (1):
- Zhongshan Hospital of Fudan University, Shanghai, Shanghai Municipality, China